CLINICAL TRIAL: NCT01057381
Title: Dose Response Relationship of Dexmedetomidine in Decreasing Post Operative Analgesic Requirements in the Pediatric Tonsillectomy Patient
Brief Title: Dexmedetomidine in Pediatric Tonsillectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Olutoyin A. Olutoye, Associate Professor of Anesthesiology & Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-17558
Record Dates: First submitted 2010-01-25; First posted 2010-01-27 (Estimated); Results first posted 2021-02-01 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Pediatric Adenotonsillectomy; Post Operative Analgesia
Keywords: Adenotonsillectomy; Postoperative analgesia; Pediatrics
MeSH Terms: interventions — Dexmedetomidine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dexmedetomidine 0.75 mcg/kg (Active Comparator): Intraoperative administration for analgesia.
  Interventions: Drug: Dexmedetomidine 0.75 mcg/kg
- Dexmedetomidine 1mcg/kg (Active Comparator): Intra-operative administration of dexmedetomidine 1 mcg/kg for analgesia
  Interventions: Drug: Dexmedetomidine 1 mcg/kg
- Morphine 50 mcg/kg (Active Comparator): Intra-operative administration of morphine 50 mcg/kg for analgesia
  Interventions: Drug: Morphine 50 mcg/kg
- Morphine 100mcg/kg (Active Comparator): Intra-operative administration of morphine 100mcg/kg for analgesia
  Interventions: Drug: Morphine 100 mcg/kg

INTERVENTIONS:
Drug: Dexmedetomidine 0.75 mcg/kg — Single intra-operative administration of dexmedetomidine 0.75 mcg/kg over 10 minutes for analgesia.
  Other Names: Precedex
  Arms: Dexmedetomidine 0.75 mcg/kg
Drug: Morphine 50 mcg/kg — Single intra-operative administration of morphine 50 mcg/kg over 10 minutes for analgesia
  Other Names: Morphine
  Arms: Morphine 50 mcg/kg
Drug: Morphine 100 mcg/kg — Single intra-operative dose of morphine 100 mcg/kg over 10 minutes for analgesia
  Other Names: Morphine
  Arms: Morphine 100mcg/kg
Drug: Dexmedetomidine 1 mcg/kg — Single intra-operative administration of dexmedetomidine 1 mcg/kg over 10 minutes for analgesia
  Other Names: Precedex
  Arms: Dexmedetomidine 1mcg/kg

SUMMARY:
The hypothesis of this study is that the administration of an intra-operative dose of dexmedetomidine will result in adequate analgesia without respiratory depression thereby resulting in an early discharge from the post anesthetic care unit following adenotonsillectomy.

DETAILED DESCRIPTION:
Dexmedetomidine, an alpha 2 agonist provides some analgesia without respiratory depression. Children undergoing tonsillectomy and adenoidectomy occasionally have episodes of respiratory obstruction in the recovery room following administration of opioids.

As dexmedetomidine provides some analgesia without respiratory depression,an intra-operative dose of dexmedetomidine may provide adequate analgesia without significant side effects thereby allowing for quick post operative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Children between ages 3 and 17 years with American Society of Anesthesiology classification 1 or 2.

Exclusion Criteria:

* Children less than 3 years
* Children with uncorrected cardiac lesions
* Children with heart block or liver impairment
* Children with American Society of Anesthesiology Class 3 or 4.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2005-08; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olutoyin A Olutoye, M.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexmedetomidine 0.75 mcg/kg | Dexmedetomidine 1mcg/kg | Morphine 50 mcg/kg | Morphine 100mcg/kg
Started | 26 | 27 | 30 | 26
Completed | 26 | 27 | 30 | 26
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine 0.75 mcg/kg | Dexmedetomidine 1mcg/kg | Morphine 50 mcg/kg | Morphine 100mcg/kg | Total
Number analyzed (Participants) | 26 | 27 | 30 | 26 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 27 | 30 | 26 | 109
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 15 | 16 | 65
  Male | 8 | 11 | 15 | 10 | 44
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 26 | 27 | 30 | 26 | 109
Duration of Surgery [Mean (Standard Deviation); unit: minutes] | 22.0 (8.4) | 21.3 (9.7) | 22.8 (7.6) | 26.0 (9.5) | 23.0 (8.9)
Duration of Anesthesia [Mean (Standard Deviation); unit: minutes] | 48.2 (19.3) | 44.7 (10.8) | 43.3 (9.7) | 49.6 (13.3) | 46.3 (13.7)

OUTCOME MEASURES:

1. Primary Outcome: Amount of Post-Operative Rescue Morphine Required for Analgesia
Time Frame: From admission to discharge from PACU, up to 1 hour
Measure: Mean (Standard Deviation); unit: ug/kg
Arm/Group | Dexmedetomidine 0.75 mcg/kg | Dexmedetomidine 1mcg/kg | Morphine 50 mcg/kg | Morphine 100mcg/kg
Number analyzed (Participants) | 26 | 27 | 30 | 26
ug/kg | 45.2 (30.8) | 37.0 (25.4) | 43.3 (23.6) | 36.5 (31.0)

2. Secondary Outcome: Morphine Rescue Doses Needed by Participants
Description: Subjects with a Children's Hospital of Eastern Ontario Pain Scale score greater than 8 received rescue morphine doses of 25 ug/kg IV at 10-minute intervals until the score was less than 8.
  Minimum and Maximum values: minimum score: 4 & maximum score: 13. The higher the score ( > 8), the greater the pain appreciated by the patient.
Time Frame: From admission to discharge from PACU, up to 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine 0.75 mcg/kg | Dexmedetomidine 1mcg/kg | Morphine 50 mcg/kg | Morphine 100mcg/kg
Number analyzed (Participants) | 26 | 27 | 30 | 26
Participants
  0 dose | 6 | 3 | 1 | 4
  1 dose | 2 | 14 | 13 | 14
  >1 dose | 18 | 10 | 16 | 8

3. Secondary Outcome: Duration of Oxygen Supplementation
Description: The subjects were then transported to the PACU with supplemental oxygen. Oxygen administration was continued after extubation until the patient was awake and could sustain room air saturations greater than 95% for 5 minutes. Duration of oxygen requirement was recorded as the time from tracheal extubation to cessation of oxygen supplementation in the PACU.
Time Frame: From admission to PACU until room air saturations greater than or equal to 95% for 5 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Dexmedetomidine 0.75 mcg/kg | Dexmedetomidine 1mcg/kg | Morphine 50 mcg/kg | Morphine 100mcg/kg
Number analyzed (Participants) | 26 | 27 | 30 | 26
minutes | 17 (11) | 19 (12) | 20 (19) | 18 (14)

4. Secondary Outcome: Time to PACU Discharge Readiness
Description: Patients were considered ready for discharge from the PACU when they attained an Aldrete score of 9 or more and were free from pain, nausea, and vomiting. Aldrete score ranges form 0 to 10 and patients greater than 8 are deemed satisfactory for discharge from the PACU
Time Frame: From admission to discharge from PACU, no time limit
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Dexmedetomidine 0.75 mcg/kg | Dexmedetomidine 1mcg/kg | Morphine 50 mcg/kg | Morphine 100mcg/kg
Number analyzed (Participants) | 26 | 27 | 30 | 26
minutes | 115 (0.04) | 116 (0.03) | 117 (0.03) | 122 (0.06)

5. Secondary Outcome: Number of Participants With Emergence Agitation
Description: Patients in the PACU who were crying, restless, disoriented, unresponsive to the parent's voice, with non-purposeful thrashing movements requiring additional personnel to prevent bodily harm, and inconsolable even after parental presence, rescue analgesia and additional measures of comfort were considered to have emergence agitation.
Time Frame: From admission to discharge from PACU, no time limit
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine 0.75 mcg/kg | Dexmedetomidine 1mcg/kg | Morphine 50 mcg/kg | Morphine 100mcg/kg
Number analyzed (Participants) | 26 | 27 | 30 | 26
Participants | 5 | 4 | 4 | 1

6. Secondary Outcome: Number of Participants With Postoperative Complications
Description: Post-operative complications including emesis, prolonged oxygen requirement or post- tonsillectomy bleed assessed up to 1 hour in PACU
Time Frame: From admission to discharge from PACU, up to 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine 0.75 mcg/kg | Dexmedetomidine 1mcg/kg | Morphine 50 mcg/kg | Morphine 100mcg/kg
Number analyzed (Participants) | 26 | 27 | 30 | 26
Participants
  Nausea | 2 | 0 | 0 | 3
  Vomiting | 0 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: Subjects were monitored from beginning of surgery until discharge from Post-Anesthetic Care Unit (PACU). There was no time limit on time monitored.
Arm/Group | Dexmedetomidine 0.75 mcg/kg | Dexmedetomidine 1mcg/kg | Morphine 50 mcg/kg | Morphine 100mcg/kg
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27 | 0/30 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27 | 0/30 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/27 | 0/30 | 0/26

LIMITATIONS AND CAVEATS:
We studied a relatively healthy patient population and excluded children with documented sleep apnea by polysomnography.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2005-06-03): https://cdn.clinicaltrials.gov/large-docs/81/NCT01057381/Prot_SAP_000.pdf